CLINICAL TRIAL: NCT01012570
Title: The Effect of Adalimumab on the Bone Microstructure in Crohn's Disease (CD) Patients
Status: Terminated | Type: Observational
Why Stopped: not enough patients enrolled
Sponsor: Gerhard Rogler (Other)
Responsible Party: Sponsor-Investigator, Gerhard Rogler, Prof.Dr.Dr. gerhard Rogler, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: HUM-07-019
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Drug: Application of Adalimumab — Adalimumab will be applied according to manufacture's instruction and official guidelines.

SUMMARY:
The investigators will study the effect of Adalimumab on the bone microstructure.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* CDAI > 220 und < 450
* Biologika naiv
* CD seit > 6 Monaten

Exclusion criteria:

* other TNF-Blocker
* Steroids > 40 mg
* Malignoma in der Anamnesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients cohort of the University Hospital Zurich
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland